CLINICAL TRIAL: NCT01385267
Title: Fetal Lung Maturation in Twin Gestations Based on Birth Order and Weight Discordance
Brief Title: Fetal Lung Maturation in Twin Gestations
Status: Completed | Type: Observational
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 08074
Record Dates: First submitted 2011-06-28; First posted 2011-06-30 (Estimated); Last update posted 2018-12-28 (Actual); Status verified 2016-09

CONDITIONS: Discordance in Lung Maturity in Diamniotic Twins

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A sample of amniotic fluid will be drawn from the amniotic sac of Twin A and Twin B. Each amniotic sac will be aspirated by the obstetrician and sent to the laboratory for determination of fetal lung maturity index and lamellar body count. Fetal lung maturity index and lamellar body count will be correlated to see if there is an association between Twin A and Twin B.
  Fetal Lung Maturity index and lamellar body count will be calculated and compared based on fetal weight, sex, zigosity, and birth order. Demographic information, maternal obstetrical and medical history, newborn/fetal data, indications for cesarean section and twin A and B outcomes will be obtained through OB Traceview or patient chart.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diamniotic twin gestations
  Interventions: Procedure: aspiration of amniotic fluid

INTERVENTIONS:
Procedure: aspiration of amniotic fluid — a sample of amniotic fluid will be drawn from the amniotic sac of Twin A and Twin B. Each amniotic sac will be aspirated by the obstetrician and sent to the laboratory for determination of fetal lung maturity index and lamellar body count.
  Other Names: diamniotic twins

SUMMARY:
Objectives:

To evaluate discordance in lung maturity in diamniotic twins based on birth order, sex and body weight. If we find discordance in fetal lung maturity in twin gestations this will change current practice of sampling only one amniotic sac for evaluation of fetal lung maturity.

DETAILED DESCRIPTION:
Objectives:

To evaluate discordance in lung maturity in diamniotic twins based on birth order, sex and body weight. If we find discordance in fetal lung maturity in twin gestations this will change current practice of sampling only one amniotic sac for evaluation of fetal lung maturity.

Hypotheses:

Lung maturation within twin pairs is weakly correlated based on presentation and estimated fetal weight.

Research Methods:

This study will be prospective cohort study of women with twin diamniotic intrauterine gestations who will be delivered at a Good Samaritan or Bethesda North Hospital. Patients will be counseled and informed consent for participation in the study will be obtained prior to enrollment in study.

At the time of Cesarean delivery or in the event of amniocenteses for FLM, a sample of amniotic fluid will be drawn from the amniotic sac of Twin A and Twin B. Each amniotic sac will be aspirated by the obstetrician and sent to the laboratory for determination of fetal lung maturity index and lamellar body count. Fetal lung maturity index and lamellar body count will be correlated to see if there is an association between Twin A and Twin B.

Fetal Lung Maturity index and lamellar body count will be calculated and compared based on fetal weight, sex, zigosity, and birth order. Demographic information, maternal obstetrical and medical history, newborn/fetal data, indications for cesarean section and twin A and B outcomes will be obtained through OB Traceview or patient chart.

Study population:

Participants will include pregnant patients, greater than 24 completed weeks with diamniotic twin gestations, at Good Samaritan and Bethesda North Hospitals. Patients will be scheduled for a cesarean section by their primary MD prior to being approached for inclusion into the study.

ELIGIBILITY:
Inclusion Criteria:

Diamniotic twin gestations

* Twenty-four completed weeks gestation with dating calculated by their sure last menstrual period or utilizing a first trimester crown rump length ultrasound.
* English Speaking
* Scheduled cesarean section by patient's primary MD

Exclusion Criteria:

* Monoamniotic twins
* Presence of gross blood in amniotic sample
* Presence of meconium amniotic fluid
* Known/diagnosed fetal or newborn anomaly
* Twin to Twin Transfusion Syndrome (TTTS)
* Vaginal delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will include pregnant patients, greater than 24 completed weeks with diamniotic twin gestations, at Good Samaritan and Bethesda North Hospitals. Patients will be scheduled for a cesarean section by their primary MD prior to being approached for inclusion into the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
FLM Index | 3 years
  FLM Index
Lamellar Body Counts | 3 years
  Lamellar Body Counts

SECONDARY OUTCOMES:
Respiratory Distress Syndrome | 3 years
  Respiratory Distress Syndrome
Transient Tachypnea in newborns | 3 years
  Transient Tachypnea in newborns
Neonatal Death | 3 years
  Neonatal Death

CONTACTS AND LOCATIONS:
Overall Officials: Donna Lambers, MD, Principal Investigator — TriHealth Inc.
Locations (1):
- Good Samaritan Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No